CLINICAL TRIAL: NCT05152862
Title: Evaluation of the Criteria and Modalities of Screening for Retinopathy of Prematurity in Two French Tertiary NICU : is a Simplification Possible ?
Brief Title: Improve Screening Criteria for Retinopathy of Prematurity in Two French Center
Acronym: DEREP3
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0053
Record Dates: First submitted 2021-11-19; First posted 2021-12-10 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2022-09

CONDITIONS: Retinopathy of Prematurity
Keywords: birth weight; gestational age; premature; retina; screening
MeSH Terms: conditions — Retinopathy of Prematurity; Birth Weight; Premature Birth | interventions — Lasers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Laser — Retinal laser photocoagulation
Procedure: Anti VEGF — Anti-VEGF intravitreous injection

SUMMARY:
The aim of the study is to assess whether a delay of the first examination can be safely considered in French population. Secondary objectives are to describe retinopathy of prematurity (ROP) in a population of premature from two French tertiary NICU and to identify co-morbidities associated with the development of severe ROP.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is a major cause of blindness and visual impairment in children worldwide. Despite a stable incidence over the last decades, improvements in neonatal care and survival of extremely premature lead to an increased screening and follow up of ROP. Retinal examination is painful and can result in clinical deterioration, it also generates significant health care costs. In this way, several studies suggest the need to optimize screening without ignoring severe ROP requiring treatment. Recently, SCREENROP in Canada and SWEDROP studies in Sweden contributed to a modification of the national screening guidelines with a reducing upper limit at 30 weeks of gestational age (GA) and a postponing of the first examination. Because of the population studied, those recommendations cannot be applicable in other countries.

Recommendations in France are to screen infants < 31 GA or 1250 g, first examination should be performed at PMA 31 in infants < 27 GA and at 4 weeks postnatal age (PNA) in infants born at 27 GA or more. Our main hypothesis is that a reduction of the screening criteria by decreasing the upper limit of the threshold at 30 GA and/or postponing the first examination is acceptable in a population of premature newborns from two French tertiary NICU. This simplification of the screening modalities could reduced the number of fundus examinations performed, while limiting risks for the patient as well as costs. This study could be a pilot study for a national multicenter trial, with the objective of revising national screening guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Infant with gestational age < 31 weeks and/or birth weight < 1250 g
* With at least one retinal examination
* holders of the parental rights informed and not objecting to the study

Exclusion Criteria:

* infants died before 28 days PNA
* infants with hydrocephaly.
* infants with significant congenital malformations or genetic abnormalities.

Ages: 0 Years to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cohort will be selected among all premature born between January 2016 and November 2020 and hospitalized in Centre Hospitalier Sud Francilien (Corbeil Essonnes 91) and Hopital Robert Debré (Paris 75).
Sampling Method: Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Number of infants with type 1 or 2 ROP found at routine screening. | Day 0
  Number

SECONDARY OUTCOMES:
Time from first retinal examination to treatment of ROP | Day 0
  days
Postnatal age / SAC at first by gestational age | Day 0
  days
Time from first retinal examination to diagnostic of severe ROP | Day 0
  days

CONTACTS AND LOCATIONS:
Overall Officials: Pauline LEROUX, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- LEROUX Pauline, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No